CLINICAL TRIAL: NCT04737694
Title: Impact of Ketone Ester Supplementation on Substrate Oxidation and Physical Performance
Brief Title: Ketone Supplements and Substrate Oxidation and Physical Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20-07HC
Record Dates: First submitted 2020-11-02; First posted 2021-02-04 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Ketosis; Glucose Metabolism
MeSH Terms: conditions — Ketosis | interventions — formic acid 4-(3-oxobutyl)phenyl ester; Glucose

STUDY DESIGN:
Intervention Model Description: Double blinded randomized crossover design
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone + Carbohydrate (Experimental): 573 mg/ kg body weight ketone ester + 110 g glucose
  Interventions: Dietary Supplement: Ketone ester
- Carbohydrate (Active Comparator): Isocaloric amount of glucose to match ketone + carbohydrate
  Interventions: Dietary Supplement: Glucose

INTERVENTIONS:
Dietary Supplement: Ketone ester — Oral ketone ester + glucose supplement
  Arms: Ketone + Carbohydrate
Dietary Supplement: Glucose — Glucose supplement
  Arms: Carbohydrate

SUMMARY:
The objective of this randomized crossover study is to examine the influence of consuming a ketone ester plus carbohydrate (KE+CHO) supplement on substrate oxidation and physical performance in 15 healthy adults. Following a 48-hr muscle glycogen normalization period, volunteers will consume either an isocaloric KE+CHO (KE: 573 mg KE/kg body mass, CHO: 110 g) or isocaloric CHO drink and complete 90-min of metabolically-matched, load carriage (~30% body mass) steady-state aerobic (~60 ± 5 % of VO2peak) exercise on a treadmill. Glucose tracers will be used to assess glucose turnover, and contribution to exogenous and plasma glucose oxidation. Serial blood draws will be collected during each trial to assess endocrine and circulating substrate responses. After steady-state exercise volunteers will complete a time to exhaustion (TTE) physical performance tests at 85% VO2peak on a treadmill. Volunteers will then be provided with food for the remainder of the day. Following a 10-hr overnight fast, volunteers will return to the laboratory and consume the same supplement (KE+CHO or CHO) as they did the previous day. Volunteers will then perform a 4-mile load carriage time trial on a treadmill. Following a minimum 7-day washout period, volunteers will return to the laboratory to complete the second arm of the study. The primary risks associated with this study include those associated with exercise, blood draws, and gastrointestinal discomfort from the KE+CHO supplement.

DETAILED DESCRIPTION:
Following an overnight (10 hour) fast, two catheters will be placed into the lower arm (one in each arm). One arm will be used for infusion of 6,6-[2H2] glucose tracer and the other will be used for blood sampling under resting and exercise conditions. Following an initial blood sample collection to determine background enrichments, a primed, continuous infusion of 6,6-[2H2] glucose will begin (prime, 82.2 µmol∙kg-1; continuous rate, 0.78 µmol∙kg-1∙min-1, Figure 1). The 6,6-[2H2] glucose will be infused for 100 min under resting fasted conditions to ensure isotopic steady-state is achieved prior to initiating exercise. Volunteers will consume either an isocaloric KE+CHO (KE: 573 mg KE/kg body mass, CHO: 110 g) or CHO drink prior to and during 90-min of metabolically-matched (~60 ± 5 % of VO2peak), steady-state load carriage (~30% body mass) exercise. Drinks will be enriched with U-13C-glucose (Cambridge Isotope Laboratory, Andover, MA, USA) to increase the isotopic enrichment well above natural levels and optimize the measurement of exogenous carbohydrate oxidation. During exercise V̇O2, V̇CO2, and HR will be measured at approximately 0, 20, 45, 60, 75, and 85 min.

After the 90-min steady-state treadmill exercise, participants will complete a TTE performance test. For volunteer safety TTE performance tests will be conducted without the additional weight from the load carriage exercise. Volunteers will be given time to stretch and warm-up on the treadmill before the TTE performance test beings. Volunteers will then run on the treadmill at a fixed speed and grade that elicits 85% of their VO2peak. The TTE performance test will be determined as the time of volitional exhaustion. Following completion of the test, a self-selected cool-down will occur. Volunteers will complete a minimum of two practice exercise sessions to ensure they are familiar with the performance test.

The following day volunteers will return to the laboratory after an overnight fast. After consuming the study drink (KE+CHO or CHO) participants will complete a self-paced 4-mile load carriage (~30% body mass) time trial on a treadmill to assess aerobic performance. Time trial performance will be assessed as the total amount of time taken to complete 4 miles. The treadmill will be set at a constant 1% grade for the entire test. Following a warm-up period, volunteers will blindly modulate treadmill speed in order to complete the distance as quickly as possible. The only feedback given will be distance covered at half mile increments. At half mile increments volunteers' rate of perceived exertion will be determined using the Borg Scale. Heart rate will be monitored throughout the time trial. Heart rate will be recorded at half mile increments. No motivation will be provided during the time trial. Participants may consume water ad libitum during the time trial. Following completion of the test, a self-selected cool-down will occur. Volunteers will complete a minimum of two practice exercise sessions to ensure they are familiar with the performance test.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 39 years
* Body mass index (BMI) < 30 kg/m2
* Routinely participate in aerobic and/or resistance exercise at least 2 days per week
* Refrain from the use of caffeine, alcohol, dietary supplements, and nicotine while consuming study diets
* Supervisor approval to participate for active duty military and federal civilian employees working within the US Army Natick Soldier Systems Center

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (i.e., kidney disease, diabetes, cardiovascular disease, etc.)
* Disease or medication (i.e., diabetes medications, statins, corticosteroids, etc) that affects macronutrient utilization and/or the ability to participate in strenuous exercise
* Allergies or intolerance to foods (including but not limited to lactose intolerance/milk allergy) to be utilized in the study or vegetarian practices
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues
* Musculoskeletal injuries that compromise the ability to exercise
* Not willing to avoid non-study exercise and foods during each of the 3 day testing periods
* Blood donation within 8 weeks of beginning the study
* Pregnant or breast feeding

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Time to exhaustion | 30 minutes
  Determine the effect of ketone esters plus carbohydrate (KE + CHO) supplementation on physical performance as determine by time to exhaustion at 85% VO2max on a treadmill compared to CHO alone
Time trial | 120 minutes
  Determine the effect of ketone esters plus carbohydrate (KE + CHO) supplementation on physical performance as determine by a self paced 4 mile time trial on a treadmill compared to CHO alone
Substrate oxidatoin | 90 minutes
  Determine the effect of KE + CHO supplementation on changes in substrate oxidation during moderate-intensity load carriage exercise compared to CHO alone.

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Margolis, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howard EE, Allen JT, Coleman JL, Small SD, Karl JP, O'Fallon KS, Margolis LM. Ketone Monoester Plus Carbohydrate Supplementation Does Not Alter Exogenous and Plasma Glucose Oxidation or Metabolic Clearance Rate During Exercise in Men Compared with Carbohydrate Alone. J Nutr. 2023 Jun;153(6):1696-1709. doi: 10.1016/j.tjnut.2023.03.002. Epub 2023 Mar 8. PMID 36893935